CLINICAL TRIAL: NCT06643377
Title: An Open-Label, Multiple-Dose Clinical Study to Evaluate the Pharmacokinetics of Enlicitide in Participants With Severe Renal Impairment
Brief Title: A Clinical Study of Enlicitide in Participants With Severe Renal Impairment (MK-0616-032)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0616-032; MK-0616-032 (Other: MSD)
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Panel A: Severe Renal Impairment (Experimental): Participants with severe renal impairment receive enlicitide once daily (QD) for 28 days.
  Interventions: Drug: Enlicitide
- Panel B: Healthy (Experimental): Healthy participants receive enlicitide QD for 28 days.
  Interventions: Drug: Enlicitide

INTERVENTIONS:
Drug: Enlicitide — Oral tablet
  Other Names: Enlicitide decanoate; MK-0616

SUMMARY:
Researchers have designed a new study medicine called enlicitide decanoate as a new way to lower the amount of low-density lipoprotein cholesterol (LDL-C) in a person's blood. Enlicitide decanoate will be called "enlicitide" from this point forward, The purpose of this study is to learn what happens to enlicitide in a person's body over time (a pharmacokinetic (PK) study). Researchers will compare what happens to enlicitide in the body when it is given to people with severe renal impairment (meaning the kidneys do not work properly) and to people who are in good health. The researchers believe that the total amount of enlicitide in a person's body measured during the 24 hours after a dose will be similar in people with severe renal impairment and in healthy people.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Body Mass Index (BMI) between 18 and 40 kg/m^2, inclusive
* On a stable dose of statin therapy; no changes to dose or type of statin therapy for at least 2 months

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History or presence of renal artery stenosis
* Had a functioning renal transplant in the past 5 years and is taking transplant medication
* History of gastrointestinal (GI) disease which might affect food and drug absorption

Panel A: Participants with Severe Renal Impairment:

- History of any illness, other than hypercholesterolemia and Renal Impairment

Panel B: Healthy Participants:

- History of clinically significant endocrine, GI, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases, other than hypercholesterolemia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration versus Time Curve from Time 0 to 24 hours (AUC0-24) of enlicitide in plasma | Pre-dose and at designated time points up to 24 hours post dose on Day 28
  AUC0-24 of enlicitide in plasma will be determined.
Maximum plasma concentration (Cmax) of enlicitide in plasma | Pre-dose and at designated time points up to 24 hours post dose on Day 28
  Cmax of enlicitide in plasma will be determined.
Time to maximum plasma concentration (Tmax) of enlicitide in plasma | Pre-dose and at designated time points up to 24 hours post dose on Day 28
  Tmax of enlicitide in plasma will be determined.
Apparent Clearance (CL/F) of enlicitide in plasma | Pre-dose and at designated time points up to 24 hours post dose on Day 28
  CL/F of enlicitide in plasma will be determined.
Apparent volume of distribution during terminal phase (Vz/F) of enlicitide in plasma | Pre-dose and at designated time points up to 24 hours post dose on Day 28
  Vz/F of enlicitide in plasma will be determined.
Number of participants who experience one or more adverse events (AEs) | Up to approximately 42 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study intervention due to an AE | Up to approximately 28 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- United States (5):
  - Velocity Clinical Research, New Smyrna Beach ( Site 0003), Edgewater, Florida
  - Velocity Clinical Research, Hallandale Beach ( Site 0006), Hallandale, Florida
  - Nature Coast Clinical Research - Inverness ( Site 0002), Inverness, Florida
  - Jacksonville Center for Clinical Research ( Site 0004), Jacksonville, Florida
  - Genesis Clinical Research, LLC ( Site 0001), Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com